CLINICAL TRIAL: NCT06603922
Title: Towards a Personalized Medicine Approach to Psychological Treatment for Psychosis
Brief Title: The Personalized Psychological Treatment for Psychosis
Acronym: PERMEPSY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Polish Academy of Sciences (Other)
Collaborators: Fundació Sant Joan de Déu (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospitals of Strasbourg (Unknown); Universitat Politècnica de Catalunya (Other); Universidad de Valparaiso (Other)
Responsible Party: Principal Investigator, Łukasz Gawęda, Associate Professor, Polish Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PerMed/V/82/PERMEPSY/2023
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Schizophrenia; Psychosis; Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: personalized medicine; psychological treatment; metacognitive training; machine learning; software platform
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: The sample will be randomized into P-MCT or classical MCT in a RCT where the user's participants (patients diagnosed with non-affective psychoses) and evaluators will be blind to the treatment condition.
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessment should be provided blind to patients' allocation (MCT vs. P-MCT). Researchers should pay attention that assessors do not learn the conditions allocation. Assessors should not discuss the content of the MCT/P-MCT sessions. At the same time, assessors should not discuss patient allocation with clinical staff. Assessors should be experienced in clinical interviews with patients suffering from psychosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized MCT (P-MCT) (Experimental): Personalized Metacognitive training
  Interventions: Behavioral: Psychological treatment (P-MCT)
- Metacognitive training (MCT) (Active Comparator): Metacognitive training
  Interventions: Behavioral: Psychological treatment (MCT)

INTERVENTIONS:
Behavioral: Psychological treatment (P-MCT) — Personalization will be performed according to the results obtained from the platform. Both the classic MCT and personalized MCT will be the same with regard to specific modules that are offered to patients. However, the personalized MCT will have personalized homeworks that target specific factors, in which patients have deficits. For instance, patients with deficits in self-esteem (based on the results from the platform) will be provided with homework addressing this aspect. We identified five domains that will be personalized: 1. self-esteem; 2. cognitive insight; 3. delusions; 4. positive symptoms; 5. completion.
  Arms: Personalized MCT (P-MCT)
Behavioral: Psychological treatment (MCT) — Metacognitive training is a cognitive approach to the treatment of positive symptoms in psychosis.
  Metacognitive training consists of ten modules referring to common cognitive issues and biases in solving problems in schizophrenia. The topics of MCT include the following: attribution blaming and taking credit (module 1), jumping to conclusions (modules 2 & 7), changing beliefs (module 3), deficits in theory of mind and social cognition (modules 4 and 6), overconfidence in (memory) errors (module 5), mood (module 8), self-esteem (9) and stigma (10).
  Each session lasts 45-60 min and follows a protocol defined in the 'Metacognitive Training for Psychosis (MCT)' manual.
  The MCT for Schizophrenia programme will be applied to the group (6-12 persons) applied by therapists in each center. The training format (online or in-person) as well as the frequency (1 or 2 times per week) will vary depending on the center.
  Arms: Metacognitive training (MCT)

SUMMARY:
The main aim of the clinical trial is to validate the Machin Learning (ML) predictive model for personalized Metacognitive Training (MCT) by comparing classic MCT to personalized MCT (P-MCT) among patients diagnosed with psychosis who had a history of delusions. More precisely, we will compare classic MCT to P-MCT in a randomized clinical trial.We expect personalised MCT treatment will see more improvement than classical MCT in outcome variables measuring treatment efficacy.

DETAILED DESCRIPTION:
This prospective study will consist of a pilot, double-blind clinical trial comparing Personalized MCT (P-MCT) to classical MCT. This pilot study will serve as a basis to validate the profiling strategy of patients and to test whether a personalized approach to psychological interventions (P-MCT) is more effective than non-personalized interventions (classical MCT).

The experimental intervention will be P-MCT. Baseline data of the patients randomized to the P-MCT and classical MCT group will be entered into the prototype platform, which will output the patient's profile and an estimate of response to MCT and the specific homeworks to be included in the intervention. MCT dedicates one session to attributional biases, two to Jumping to Conclusions Bias, one to belief change, two to empathy, one to meta-memory, and one to self-esteem and two additional for self-esteem and stigma. The personalized MCT will have personalized homeworks that target specific factors, in which patients have deficits. For instance, patients with deficits in self-esteem (based on the results from the platform) will be provided with homework addressing this aspect. We identified five domains that will be personalized: 1. self-esteem; 2. cognitive insight; 3. delusions; 4. positive symptoms; 5. completion.

All interventions will be conducted by psychologists or mental-health professionals trained in MCT. All the treatments will be conducted on-site and online. Both conditions patients will receive 10 sessions of MCT. Control intervention: The control group is an active group that will receive classical MCT for psychosis following the current program. Duration of intervention per patient: 10 weeks (1 session per week of one hour of length). Patients will be assessed at baseline, post-treatment, and 6-month follow up.

The sample will include patients with Schizophrenia Spectrum Disorders (n=252) from five clinical center (Poland, Germany, France, Chile and Spain).

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients and outpatients with a DSM-IV-R and DSM-5 diagnosis of non-affective psychosis or Clinical High Risk for psychosis.
2. Presence of positive symptoms during the last year (PANSS delusions, suspiciousness or grandiosity >=3).
3. Adults, 18 - 65 years of age
4. Stable condition with no expected changes in medication (information from clinical services).
5. Lack of severe cognitive deficits (global assessment or/and information from clinical services);

Exclusion Criteria:

1. Having received MCT in the previous year.
2. Neurological disorder, a history of head trauma or premorbid IQ below 70 (based on medical reports and/or other sources);
3. A score above 5 in the "Hostility" and the "Suspiciousness" items of the PANSS Positive subscale (to preserve group dynamics).
4. aggressive behavior (reports from clinical services if available)
5. High risk of suicide (verified with DIAMOND)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic Questionnaire | Baseline
  A sociodemographic sheet will be captured the following information: age, gender/sex, marital status, years of education, living situation, number of siblings, whether they live in rural or urban areas, employment status, symptom onset, previous hospitalisations, history of suicide attempts, family mental health history, current substance use, current pharmacological treatment (name and dosage), diagnosis (options: schizophrenia,unspecified psychotic disorder, schzoaffective disorder, delusional disorder, brief psychotic disorder, schizophreniform disorder), comorbidity, other medical illnesses, and in female patients, age at menarche, age at menopause, hormone treatment (if applicable), menstrual cycle description, date of last menstrual period, amenorrhoea.
PSYRATS | baseline, post-treatment and 6-month follow-up
  Psychotic Symptom Rating Scale. The PSYRATS comprises hallucinations (11 items) and delusions (6 items) subscales, each one designed to assess the psychological aspects of the symptoms on a five-point scale, from 0 to 4.
PANSS | baseline, post-treatment and 6-month follow-up
  The Positive and Negative Syndromes Scale.PANSS is a semi-structured interview assessing 30 symptoms on a 7-point scale, from 1 (absent) to 7 (extreme). Symptoms are rated over seven days prior to the assessment.
RSES | baseline, post-treatment and 6-month follow-up
  Rosenberg's Self-Esteem Scale.A 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. The scale is believed to be unidimensional. All items are answered using a 4-point Likert scale ranging from strongly agree to strongly disagree.
BCIS | baseline, post-treatment and 6-month follow-up
  Beck Cognitive Insight Scale.The BCIS aims to assess patients' self-reflectiveness about cognitive processes and problems and (over-) confidence in decision-making. The self-report questionnaire consists of 15 items which measure "self-reflectiveness" (9 items; e.g., "At times, I have misunderstood other people's attitudes towards me.") and "self-certainty" (6 items; e.g., "My interpretations of my experiences are definitely right."). A composite index of the BCIS termed "cognitive insight" is calculated by subtracting the self-certainty subscore from the self-reflectiveness subscore.

SECONDARY OUTCOMES:
GAF | baseline, post-treatment and 6-month follow-up
  Global Assessment of Functioning. A numeric scale used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of an individual, i.e., how well one is meeting various problems in living. Scores range from 100 (extremely high functioning) to 1 (severely impaired).
DIAMOND | baseline
  structured clinical interview that queries the DSM-5 diagnostic criteria
WHOQOL-BREF | baseline, post-treatment and 6-month follow-up
  The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale.
TEC | baseline
  Traumatic Experience Checklist. The TEC is a self-report measure addressing 29 types of potentially traumatic events. It is a 29-item retrospective self-report scale. It is a reliable and valid self-report instrument that can be used in clinical practice and research. Different scores can be calculated, including a cumulative score, and scores for emotional neglect, emotional abuse, physical abuse, sexual harassment, sexual abuse, and bodily threat from a person. Only 19-item will be used.
CBQp | baseline, post-treatment and 6-month follow-up
  The CBQp is a 30-item questionnaire designed to assess cognitive biases. The questionnaire presents situations frequently encountered in everyday life, along with three response choices reflecting what an individual might think in these situations. The subscales are meant to measure: Internationalising, Catastrophizing, Jumping to Conclusions, Dichotomous Thinking, and Emotional Reasoning biases. In addition, the questions were inspired by two themes relating to psychosis: Anomalous Perceptions (AP) and Threatening Event (TE). A 13-item version of the CBQ will be used.
ISMI | baseline, post-treatment and 6-month follow-up
  Brief version of the Internalized Stigma of Mental Illness Scale. The original ISMI scale is a 29-item questionnaire designed to measure the subjective experience of stigma. Each item is rated on a four-point Likert scale from 1 (strongly disagree) to 4 (strongly agree). The subscales measure: Alienation, Stereotype Endorsement, Perceived Discrimination, Social Withdrawal, and Stigma Resistance. A 10-item version of the ISMI containing the two strongest items from each subscale.
QSLE-SV | baseline, post-treatment and 6-month follow-up
  Short version of the questionnaire of stressful life events. The original QSLE scale is a 52-item questionnaire designed to measure stressful life events. The abbreviated QSLE-SV with 18 items shows the importance of different life dimensions such as education, work, family, legal and health. In the study, we will use 9 items from the abbreviated version of the tool.
RFQ | baseline, post-treatment and 6-month follow-up
  The Reflective Functioning Questionnaire. The RFQ is a brief 8-item self-report measure of mentalizing, i.e., the capacity to interpret the self and others in terms of internal mental states such as feelings, wishes, goals, desires, and attitudes. Individuals in the RFQ respond to each item on a seven-point scale between "strongly disagree" and "strongly agree" response options.
ISI | baseline, post-treatment and 6-month follow-up
  Insomnia Severity Index. The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. The usual recall period is the "last two weeks" and the dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28.
SUMD | baseline, post-treatment and 6-month follow-up
  The Scale to Assess Unawareness of Mental Disorder. The SUMD is a 20-item scale that assesses current and past awareness of illness. The first three items, which assess general awareness of mental illness, are (1) awareness of mental disorder, (2) effects of medication, and (3) social consequences of mental disorder. Items 4-20 pertain to specific symptoms. If the subject shows awareness of a symptom, he/she is asked about the attribution of this symptom. Awareness and attribution items are rated from 1 to 5, with higher scores indicating poorer awareness or attribution. The 17 symptom items render four subscale scores: current awareness, past awareness, current attribution, and past attribution. Only 3-item of SUMD will be used.
B-IRI | baseline, post-treatment and 6-month follow-up
  Brief Form of the Interpersonal Reactivity Index. The IRI is designed to measure empathy as a set of constructs in addition to a unitary concept. The 28-item IRI is a self-report measure consisting of four 7-item subscales: Perspective Taking (tendency to adopt the psychological point of view of others); Fantasy (tendency to transpose oneself imaginatively into the feelings and actions of fictitious characters in books, movies, and plays); Empathic Concern (feelings of sympathy and concern for others); and Personal Distress (feelings "self-oriented" feelings of personal anxiety and unease in tense interpersonal settings). B-IRI is a short version of IRI containing a 16-item scale.
BHS | baseline, post-treatment and 6-month follow-up
  Short Version of the Beck Hopelessness. The original BHS is a 20-item self-report inventory designed to measure three major aspects of hopelessness: feelings about the future, loss of motivation, and expectations. It is a true-false test that measures the extent of the respondent's negative attitudes, or pessimism about the future. It may be used as an indicator of suicidal risk in depressed people who have made suicide attempts. The short version of BHS is a 4-item scale, which includes all the affective, cognitive, and motivational components of hopelessness.
PHQ-9 | baseline, post-treatment and 6-month follow-up
  The Patient Health Questionnaire-9. The PHQ-9 is the 9-item depression module from the full PHQ. As a severity measure, the PHQ-9 score can range from 0 to 27, since each of the nine items can be scored from 0 (not at all) to 3 (nearly every day).
IPSAQ | baseline, post-treatment and 6-month follow-up
  The Internal, Personal, and Situational Attributions Questionnaire. The IPSAQ has 32 items describing 16 positive and 16 negative social situations in the second person. For positive and negative events two measures of internality are derived from responses: a measure of self-blame and a measure of the extent to which external attributions implicate others as opposed to situations. Three positive and three negative subscale scores are generated by summing the number of internal attributions, the number of personal attributions and situational attributions chosen for both the positive and negative items. Two cognitive bias scores are derived from these six subscale scores (External and Personalizing bias). We will use 4 items - 2 positive and 2 negative situations
Satisfaction with MCT treatment | post-treatment
  A questionnaire evaluating subjective training success will be handed out to the patients at the end of the training. This subjective appraisal rating was previously used in a study on the MCT (Moritz and Woodward, 2007), which found the internal consistency to be satisfactory (Cronbach's alpha = .73). The measure contained ten items covering distinct aspects of training satisfaction: effectiveness, usefulness, applicability to daily life, transparency of the aims and fun. Each item had to be rated on a 5-point scale (1 = does not agree at all - 5 = totally agree). Higher scores thus designated greater satisfaction.
TMT | baseline, post-treatment and 6-month follow-up
  The Trail-Making Test. The TMT is a neuropsychological test that involves visual scanning and working memory. The TMT has two parts: the TMT-A (rote memory) and TMT-B (executive functioning). In each test, the participant is asked to draw a line between 24 consecutive circles randomly arranged on a page. The TMT-A uses all numbers, whereas the TMT-B alternates numbers and letters, requiring the patient to switch between numbers and letters in consecutive order. The TMT is scored by how long it takes to complete the test. The time includes the correction of errors prompted by the examiner. If the person cannot complete the test in 5 minutes, the test is discontinued.
Fish Task | baseline, post-treatment and 6-month follow-up
  he Fish Task is a computerized variant of the probabilistic reasoning task designed to capture jumping to conclusion, a prominent bias targeted by two modules of MCT.
BCFT | baseline, post-treatment and 6-month follow-up
  Baron Cohen's Face Test. Facial emotion recognition test originally developed in the construction of the Reading the Mind in the Eyes Test. BCFT consists of 20-items showing pictures of an actress displaying an emotion.Participants must choose which emotion the actress is feeling between two different choices of response. Half of the items display basic emotions, whilst the other half displays complex mental states. We will use a 4-item version and additionally participants will be asked for their confidence rated on a 5-point scale.
The Hinting Task | baseline, post-treatment and 6-month follow-up
  This task is a measure of the ability to infer the 'real intentions' behind indirect comments. It consists of 10 short passages, each describing a social interaction between two characters, ending with one character 'dropping' a hint to the other. Subjects were required to infer the actual meaning of the hint. If a subject fails to give a correct answer, a more obvious hint is provided. An appropriate response to the first hint is scored with two points. If a correct response is given only after a more obvious hint, a score of one was given. If the subject fails to give a correct answer to either of the two hints, a score of zero was given. A random selection of three stories will be presented to participants.
Monitoring symptoms during MCT | post-treatment
  After every session, participants will receive a brief questionnaire assessing the severity of the present symptoms (cognitive biases - 4 items (based on DACOBS, Davos Assessment of the Cognitive Biases Scale), positive symptoms - 4 items, negative/affective symptoms - 6 items (basen on PRISS, Patient-Reported Impact of Symptoms in Schizophrenia Scale ).

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Gawęda, Professor, Principal Investigator — The Institute of Psychology, Polish Academy of Sciences
Locations (6):
- Universidad de Valparaíso, Valparaíso, Región de Valparaíso, Chile
- University Hospitals of Strasbourg, Strasbourg, Strasbourg Cedex, France
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany
- The Institute of Psychology, The Polish Academy of Sciences, Warsaw, Warsaw, Poland
- Spain (2):
  - Fundació Sant Joan de Déu, Barcelona, Barcelona
  - Universitat Politècnica de Catalunya, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: No